CLINICAL TRIAL: NCT01682018
Title: Clinical Trial to Evaluate the Value of Bronchoscopic Lung Volume Reduction by Endobronchial Valves in Patients With Single Lung Transplantation and Overinflation of the Native Lung
Brief Title: The Value of Bronchoscopic Lung Volume Reduction by Endobronchial Valves in Patients With Single Lung Transplantation and Overinflation of the Native Lung
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC126908
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-07

CONDITIONS: Native Lung Overinflation in Patients That Underwent Single Lung Transplantation Due to Emphysema
Keywords: emphysema; lung transplantation
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention group (Experimental): Patients that underwent dingle lung transplantation due to emphysema and developed native lung overinflation as demonstrated by chest CT and decline in pulmonary lung function tests (FEV1 ) shall undergo valves placement to the native lung
  Interventions: Device: lung volume reduction using the Zephyr device

INTERVENTIONS:
Device: lung volume reduction using the Zephyr device — lung volume reduction using the Zephyr device

SUMMARY:
The purpose of the study is to investigate if bronchoscopic lung volume reduction by valves (Zephyr) would reduce native lung overinflation in patients that underwent single lung transplantation due to emphysema, and improve their well being and pulmonary function tests.

DETAILED DESCRIPTION:
Emphysema is a progressive pulmonary disease characterized by abnormal and permanent enlargement of air spaces distal to terminal bronchioles accompanied by the destruction of pulmonary parenchyma. Treatment includes inhaled bronchodilator therapy, rehabilitation and/or oxygen treatment. In addition to the above, patients with severe emphysema may benefit from surgical lung volume reduction and/or lung transplantation. The rationale for lung volume reduction surgery is that reducing lung size would restore elastic recoil of the lung and improve chest wall and diaphragm mechanics. It has previously been shown that particularly patients with heterogeneous emphysema seem to benefit most from surgical lung volume reduction.

Bronchoscopic lung volume reduction (BLVR) has recently been introduced as a less invasive potential alternative to surgical lung volume reduction. BLVR attempts to achieve the effects of surgery, by placing bronchial prostheses using a fibreoptic bronchoscope to selectively occlude the airways supplying the most affected hyperinflated regions of the emphysematous lung, while permitting exhaled gas to escape. This attempts to achieve segmental or lobar volume reduction, simulating the effects of surgical LVR.

The purpose of the study is to investigate if bronchoscopic lung volume reduction by valves (Zephyr) would reduce native lung overinflation in patients that underwent single lung transplantation due to emphysema, and improve their well being and pulmonary function tests

ELIGIBILITY:
Inclusion Criteria:

Single lung transplantation due to emphysema at least six months following transplantation that developed native lung overinflation

* Age from 40 to 75 years
* BMI < 32 kg/m2
* FEV1 < 40% of predicted value, FEV1/FVC < 70%
* TLC > 120% predicted, RV > 150% predicted.
* Stable with < 20 mg prednisone (or equivalent) qd
* PaCO2 < 50mm Hg
* PaO2 > 45 mm Hg on room air
* 6-min walk of > 50m (without rehabilitation) or > 100m (with rehabilitation)
* Nonsmoking for 4 months prior to initial interview and throughout screening
* The patient agrees to all protocol required follow-up intervals.
* The patient has no child bearing potential
* The patient is willing and able to complete protocol required baseline assessments and procedures Exclusion criteria
* Prior endobronchial treatment for emphysema
* Pleural or interstitial disease that precludes surgery.
* Prior lung transplant, LVRS, median sternotomy, bullectomy or lobectomy.
* Clinically significant bronchiectasis
* Pulmonary nodule requiring surgery
* History of recurrent respiratory infections (> 3 hospitalization in the last year)
* Clinically significant (> 4 Tablespoons per day) sputum production
* Fever, elevated white cell count, or other evidence of active infection
* Dysrhythmia that might pose a risk during exercise or training
* Congestive heart failure within 6 mo and LVEF < 45%
* Evidence or history of Cor Pulmonale
* Resting bradycardia (< 50 beats/min), frequent multifocal PVCs, complex ventricular arrhythmia, sustained SVT
* History of exercise-related syncope
* MI within 6 mo and LVEF < 45%
* Evidence of systemic disease or neoplasia expected to compromise survival during 5-yr period
* Any disease or condition that interferes with completion of initial or follow-up assessments
* Patient is currently enrolled in another clinical trial
* Patient is unable to complete 3 minutes of unloaded peddling on cycle ergometer
* Alpha-1-Antitrypsin Deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
•Mean % change in lung function (FEV1) | 90 days

SECONDARY OUTCOMES:
Mean change in six minutes walk distance | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel, Israel